CLINICAL TRIAL: NCT05892393
Title: Pilot PET Imaging Study of [89Zr]DFO-YS5 for Detecting CD46 Positive Malignancy in Multiple Myeloma
Brief Title: Imaging Study of [89Zr]DFO-YS5 for Detecting CD46 Positive Malignancy in Multiple Myeloma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Robert Flavell, MD, PhD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Robert Flavell, MD, PhD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23925; NCI-2023-04068 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); R01CA271606 (NIH)
Record Dates: First submitted 2023-05-26; First posted 2023-06-07 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma; Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A ([89Zr]DFO-YS5, single scan (Experimental): Participants receive [89Zr]DFO-YS5 IV and undergo a single PET/CT or PET/MRI scan 5-7 days post-injection. Participants also receive fludeoxyglucose F-18 IV and undergo PET/CT or PET/MRI scan within 28 days prior to day 1
  Interventions: Drug: Zirconium Zr 89-DFO-YS5; Procedure: Positron Emission Tomography / Computed Tomography (PET/CT); Procedure: Positron Emission Tomography / Magnetic Resonance Imaging (PET/MRI); Other: Fludeoxyglucose F-18
- Cohort B ([89Zr]DFO-YS5, multiple scans (Experimental): Participants receive [89Zr]DFO-YS5 IV and undergo four PET/CT or PET/MRI scans on days 1, 2, 3-4, and 5-7 post-injection. Participants also receive fludeoxyglucose F-18 IV and undergo PET/CT or PET/MRI scan within 28 days prior to day 1
  Interventions: Drug: Zirconium Zr 89-DFO-YS5; Procedure: Positron Emission Tomography / Computed Tomography (PET/CT); Procedure: Positron Emission Tomography / Magnetic Resonance Imaging (PET/MRI); Other: Fludeoxyglucose F-18

INTERVENTIONS:
Drug: Zirconium Zr 89-DFO-YS5 — Given IV
  Other Names: (89)Zr-DFO-YS5; 89Zr DFO-YS5
Procedure: Positron Emission Tomography / Computed Tomography (PET/CT) — Positron emission tomography-computed tomography is a nuclear medicine technique which combines, in a single gantry, a positron emission tomography scanner and an x-ray computed tomography scanner, to acquire sequential images from both devices in the same session, which are combined into a single superposed image
  Other Names: PET/CT
Procedure: Positron Emission Tomography / Magnetic Resonance Imaging (PET/MRI) — Positron emission tomography-magnetic resonance imaging is a hybrid imaging technology that incorporates magnetic resonance imaging soft tissue morphological imaging and positron emission tomography functional imaging.
  Other Names: PET/MRI
Other: Fludeoxyglucose F-18 — Given IV
  Other Names: Fludeoxyglucose (18F)

SUMMARY:
This phase I trial tests the safety of [89Zr]DFO-YS5 positron emission tomography (PET) imaging and how well it works to detect CD46 positive cancer cells in patients with multiple myeloma. [89Zr]DFO-YS5 is an imaging agent called a radiopharmaceutical tracer. A radiopharmaceutical tracer uses a small amount of radioactive material that is injected into a vein to help image different areas of the body. [89Zr]DFO-YS5 targets a specialized protein called CD46, which is in certain multiple myeloma cancer cells, and [89Zr]DFO-YS5 PET scans may improve detection of multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the sensitivity of metastatic lesion detection in multiple myeloma using zirconium Zr 89-DFO-YS5 ([89Zr]DFO-YS5 PET, as compared with fludeoxyglucose F-18 (18F-FDG) PET imaging.

SECONDARY OBJECTIVES:

I. To determine the safety of [89Zr]DFO-YS5. II. To determine the average organ uptake of [89Zr]DFO-YS5. III. To descriptively report the patterns of intra-tumoral uptake of [89Zr]DFO-YS5 on whole body PET, including by site of disease, uptake by tumor type, inter-tumoral and inter-patient heterogeneity, and tumor-to-background signal.

IV. To calculate the dosimetry of [89Zr]DFO-YS5 in patients with multiple myeloma.

EXPLORATORY OBJECTIVE:

I. To determine the association between uptake (standardized uptake value maximum [SUVmax]) of [89Zr]DFO-YS5 with 1q amplification by fluorescence in situ hybridization (FISH) on tumor biopsies (when available; FISH may be conducted as part of routine, standard-of-care).

OUTLINE: Participants are assigned to 1 of 2 cohorts based on participant preference.

COHORT A: Participants receive [89Zr]DFO-YS5 intravenously (IV) and undergo a single PET/CT or PET/MRI scan 5-7 days post-injection. Participants also receive fludeoxyglucose F-18 IV and undergo PET/CT or PET/MRI scan within 28 days prior to day 1.

COHORT B: Participants receive [89Zr]DFO-YS5 IV and undergo four PET/CT or PET/MRI scans on days 1, 2, 3-4, and 5-7 post-injection. Participants also receive fludeoxyglucose F-18 IV and undergo PET/CT or PET/MRI scan within 28 days prior to day 1.

Patients are followed up at 30 days after final scan.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed multiple myeloma by International Myeloma Working Group (IMWG) diagnostic criteria
* At least one positive myelomatous lesion found on 18F-FDG PET/CT or PET/MRI. A positive lesion is defined as uptake greater than liver on FDG PET, based on the Italian myeloma criteria for PET use (IMPeTUs) criteria
* Age >= 18 years
* Total bilirubin =< 1.5 X institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) =< 3 X ULN
* Alanine aminotransferase (ALT) =< 3 X ULN
* Creatinine clearance >= 60 mL/min, calculated using the Cockcroft-Gault equation or serum creatinine <= 1.5x the institutional upper limit of normal.
* Ability to understand a written informed consent document, and the willingness to sign it

Exclusion Criteria:

* Any condition that, in the opinion of the principal investigator, would impair the participants' ability to comply with study procedures or interfere with the safety of the investigational regimen
* Individuals who are pregnant or breastfeeding/chestfeeding.
* - Breast-feeding/chest-feeding should be discontinued before administration of [89ZR]DFO-YS5.
* Females of childbearing potential must have a negative urine or serum pregnancy test (i.e., human chorionic gonadotropin test) within 72 hours prior to administration of [89ZR]-DFO-YS5.
* - If the urine pregnancy test is positive or equivocal, a confirmatory serum pregnancy test is required. In such cases, the individual must be excluded from participation if the serum pregnancy result is positive.
* - A female is considered to be of childbearing potential (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice), unless it is documented that the individual meets either of the following two criteria: (1) has reached a postmenopausal state ( >= 12 continuous months of amenorrhea with no identified cause other than menopause); or (2) has undergone surgical sterilization (i.e., hysterectomy and/or bilateral oophorectomy for removal of uterus and/or ovaries).
* Individuals who are pregnant or breastfeeding/chestfeeding are excluded because there is an unknown but potential risk for adverse effects in the unborn/nursing child secondary to treatment of the study participant with [89ZR]-DFO-YS5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of metastatic lesion | Up to 1 week
  Defined as the rate of lesions with positive uptake when compared against 18F-fluorodeoxyglucose (FDG) PET/computed tomography (CT) positivity. Sensitivity estimated based on lesion level without considering the location of the lesions or the possible intracorrelation of the lesions from the same patient by point estimate with its 95% confidence interval.
Median maximum standardized uptake value (SUVmax) | Up to 1 week
  The median and range of standardized uptake value maximum (SUVmax) (across all metastatic lesions per participant) in each study cohort will be descriptively reported using mediastinal blood pool and normal organ background uptake values.
Median Standardized Uptake Value averaged across lesions (SUVmax-avg) | Up to 1 week
  The median and range of SUVmax-average across all lesions in each study cohort will be descriptively reported using mediastinal blood pool and normal organ background uptake values.

SECONDARY OUTCOMES:
Proportion of participants reporting treatment-related Adverse Events | Up to 35 days
  Will be reported descriptively using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Average organ uptake of [89Zr]DFO-YS5 | Up to 1 week
  Regions of interest will be drawn on major organs, and the SUVmax calculated for each patient. Average organ uptake reported with descriptive statistics, including the mean and standard deviation (SD).
Descriptive patterns of intra-tumoral uptake of [89Zr]DFO-YS5 | Up to 1 week
  On whole body PET, site of disease, uptake by tumor type, inter-tumoral and inter-patient heterogeneity, and tumor-to-background signal. The median and range for intra-tumoral SUVmax within metastatic lesions will be reported descriptively on a per-lesion basis to assess for intra-tumoral heterogeneity and differences in uptake by site of disease.
Dosimetry measurements (Cohort B only) | Up to 1 week
  Dosimetry calculations will be performed and reported in millisievert (mSv)/megabecquerels (MBq) on a per-patient basis. Time-activity curves will be generated for each organ, and curve-fitting will be performed to derive the time-integrated activity coefficients

CONTACTS AND LOCATIONS:
Overall Officials: Robert Flavell, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No